CLINICAL TRIAL: NCT06865820
Title: Implementation and Cost Evaluation of Project UPLIFT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ngoc Cam Escoffery, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00008582; CDC-STUDY00008582 (Other: Centers for Disease Control and Prevention)
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Project UPLIFT (Experimental): Adults with epilepsy participating in a group-based program for 8 weeks. Project UPLIFT is designed to increase knowledge and skills, decrease depressive symptoms and improve quality of life.
  Interventions: Behavioral: Project UPLIFT

INTERVENTIONS:
Behavioral: Project UPLIFT — Project UPLIFT is a Mindfulness-based Cognitive Behavioral Therapy program teaching participants methods that include challenging thoughts, behavioral activation, coping, problem-solving, and mindfulness. The program is group-based and provides weekly sessions, delivered remotely via telephone or video conferencing platform, over an 8-week period.

SUMMARY:
This study tests Project Using Practice and Learning to Increase Favorable Thoughts (UPLIFT) which is a Mindfulness-based Cognitive Behavioral Therapy program teaching participants with epilepsy methods that include challenging thoughts, behavioral activation, coping, problem-solving, and mindfulness, for well-being and costs. Project UPLIFT is delivered as weekly sessions over 8 weeks.

DETAILED DESCRIPTION:
Over 3.4 million people in the US have epilepsy, which is a chronic neurological condition that affects individuals across their lifespan. A key feature of epilepsy is the unpredictable occurrence of seizures that can have catastrophic physical and psychological consequences. Even when seizures are well-controlled with anti-seizure medications (ASMs), challenges often persist leading to increased morbidity, mortality, and a decreased quality of life (QOL). Individuals with epilepsy often deal with a complex set of medical and psychosocial issues including stigma and social isolation resulting from misconceptions about epilepsy, lack of understanding around the abilities of people with epilepsy, and a fear of seizures in general. Comorbidities such as cognitive impairment and depression are common in people with epilepsy irrespective of age, gender, and socioeconomic status and are often more disabling than the seizures. Risk factors for poor outcomes in epilepsy include ASM non-adherence and poor social supports, and racial and ethnic minorities and individuals of lower socioeconomic status are particularly likely to have epilepsy complications and poor QOL.

Epilepsy also imposes a substantial economic burden on the individuals impacted, their families, and society. Costs associated with epilepsy illustrate the complexity and financial burden of the disease on the individual and system. A recent study, estimating the prevalence of and characterized health care spending for persons classified with seizure or epilepsy using 2010-2018 Medical Expenditure Panel Survey (MEPS) data across the United States determined direct health care spending for the 3.4 million community dwelling individuals with epilepsy and seizures was approximately $24.5 billion annually over the period 2010-2018; and spending for epilepsy and/or seizures is rising at approximately twice the rate as overall health care spending.

For over 17 years, the Managing Epilepsy Well (MEW) Network has provided evidence and research addressing comorbidities and other epilepsy related challenges. It was created in 2007 with support from the Centers of Disease Control and Prevention (CDC) and the CDC Epilepsy Program. One of the epilepsy self-management programs that has been developed, tested, and deemed evidence-based is Project Using Practice and Learning to Increase Favorable Thoughts (UPLIFT). Project UPLIFT focuses on depressive symptoms.

For persons with epilepsy (PWE), self-management specifically includes medication adherence, learning more about their seizures and diagnosis, keeping a seizure diary, or tracking seizures, understanding and avoiding seizure triggers, and reducing stressors that may induce a seizure. The Institute of Medicine's critical goal of epilepsy education identifies three categories of epilepsy self-management, including medication management, behavior changes to help manage epilepsy, and emotional support for dealing with a chronic condition. Epilepsy self-management programs are low-cost, manualized, and designed to overcome transportation barriers-and yet they are not utilized at their fullest potential due to barriers such as limited resources for program adoption, bias in the medical community, and information deficits about efficacy, program delivery, and costs.

Project UPLIFT is a group-based program designed to help increase knowledge and skills, reduce depressive symptoms, and improve quality of life. All study participants will receive the UPLIFT program which is provided as a weekly session over an 8-week period. The study design is a quasi-experimental pretest, posttest evaluation study with a follow-up period of up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older
* Diagnosis of epilepsy (self-reported by patient)
* Can speak English
* Has access to a phone or computer

Exclusion Criteria:

* Inability to cognitively participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-8) Score | Baseline, Month 3, Month 6
  The effectiveness of Project UPLIFT is assessed by examining depressive symptoms. The Patient Health Questionnaire (PHQ-8) is an 8-item instrument asking how often respondents have been bothered by certain problems over the past two weeks. Responses are given on a 4-point scale where "not at all" = 0 and "nearly every day" = 3. Total scores range from 0 to 24 where higher scores indicate increased symptoms of depression.
Quality of Life in Epilepsy (QOLIE-10) Score | Baseline, Month 3, Month 6
  The effectiveness of Project UPLIFT is assessed by examining quality of life. The Quality of Life in Epilepsy (QOLIE-10) instrument has 10 questions about health and daily activities. Responses are given on a range of scales, from 1 (the most positive quality of life) to 4 or 6 (the most negative quality of life). Some items are reverse scored. The final score is the average of scores for the individual items. Lower scores indicate greater quality of life while higher scores indicate greater problems from epilepsy.
Quality of Patient-Reported Outcomes Measurement Information System (PROMIS): PROMIS-Preference (PROPr) Score | Baseline, Month 3, Month 6
  The effectiveness of Project UPLIFT is assessed by examining health utility. The PROMIS-Preference (PROPr) focuses on 7 PROMIS domains of: Cognitive Function - Abilities; Depression; Fatigue; Pain Interference; Physical Function; Sleep Disturbance; and Ability to Participate in Social Roles and Activities. The PROPr scoring system has single-attribute scoring functions and a multiplicative multi-attribute scoring function for the 7 PROMIS domains. For the single-attribute scoring functions, 0 = the unhealthiest level of the domain and the healthiest levels on all other domains (disutility of the domain under examination), while 1 = utility of full health. For the multi-attribute scoring function, 0 = the utility of dead, and 1 = the utility of full health.

SECONDARY OUTCOMES:
Global Assessment of Severity of Epilepsy (GASE) Scale Score | Baseline, Month 3, Month 6
  The effectiveness of Project UPLIFT is assessed by examining seizure severity. Seizure severity is assessed with the Global Assessment of Severity of Epilepsy (GASE) Scale. The GASE is a single-item instrument completed by clinicians to rate the overall severity of the individual's epilepsy. Responses range from 1 = "not at all severe" to 7 = "extremely severe."

CONTACTS AND LOCATIONS:
Overall Officials: Cam Escoffery, PhD, MPH, Principal Investigator — Emory University; Katie Bullinger, MD, PhD, Principal Investigator — Emory University; Robin McGee, PhD, MPH, Principal Investigator — Emory University; David H Howard, PhD, Principal Investigator — Emory University
Locations (1):
- Rollins School of Public Health, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data collected before and after the intervention will be made available for sharing with other researchers.
Supporting Information: Study Protocol, SAP
Time Frame: Individual participant data will be made available for sharing immediately following publication(s) of this study.
Access Criteria: Data will be available for sharing with researchers who provide sound research questions and a sound proposal, in order to achieve aims of the proposal. Data will be available on Emory Dataverse. Researchers interested in sharing this data can contact the study PI at cescoff@emory.edu.